CLINICAL TRIAL: NCT01555879
Title: Abatacept in T3: A Characterization of Abatacept's Efficacy and Outcomes From a Real-Word Clinical Practice Information Hub on Novel Patient Sub-Groups
Brief Title: Real-world Clinical Efficacy of Abatacept in the T3 Data Registry
Status: Completed | Type: Observational
Sponsor: Arthritis Northwest PLLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-322; ANW_20110816 (Other: Arthritis Northwest)
Record Dates: First submitted 2012-02-29; First posted 2012-03-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Retrospective; Database; Data warehouse; Data mining; Collaborative effectiveness; Comparative effectiveness; Outcome based medicine; Evidence based medicine
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients in T3 who have used Abatacept for at least 3 months between 2009-03-17 and 2011-11-30.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — As prescribed by a doctor for patient medical care.
  Other Names: Orencia Intravenous

SUMMARY:
The purpose of this study is to assess the effectiveness of Abatacept in real-world clinical practice. The main hypothesis to be examined in this study is, "Abatacept's effectiveness results in a single real-world clinic (n = 100) are reproducible at another site (n ~= 200)".

DETAILED DESCRIPTION:
Two secondary hypotheses that will be tested are:

* Abatacept aids in achieving low disease activity or clinical remission in patients of the following Rheumatoid Arthritis (RA) sub-groups: RF+/CCP+, RF+/CCP- RF-/CCP+ RF-/CCP-; first time on a bio-tech drug; having previously failed a biological drug; having interstitial lung disease; identified as disabled; twenty-eight individual joints identified as {swollen, painful, tender, deformed or having decreased range of motion}; on or not on oral DMARD; age; or gender.
* A database with sufficient attributes exists from which a patient's efficacy on abatacept is accurately predictable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis
* Have used Abatacept for 3 or more months

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All rheumatoid arthritis patients from a single site who have been on Abatacept for greater than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of abatacept by analyzing the change in CDAI, DAS28, and RAPID3 scores. | Change from baseline in CDAI, DAS28, and RAPID3 scores at approximately 6 months.

SECONDARY OUTCOMES:
Determine the efficacy of abatacept by analyzing the change in CDAI, DAS28, and RAPID3 scores. | Change from baseline in CDAI, DAS28, and RAPID3 scores at approximately 3 months.
Determine the efficacy of abatacept by analyzing the change in CDAI, DAS28, and RAPID3 scores. | Change from baseline in CDAI, DAS28, and RAPID3 scores at approximately 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Knapp, Ph.D., Study Director — Arthritis Northwest PLLC; Gary Craig, M.D., Principal Investigator — Arthritis Northwest PLLC
Locations (1):
- Arthritis Northwest, Spokane, Washington, United States

REFERENCES:
- [Background] Michael Schiff, Coralie Poncet, and Manuela Le Bars International Journal of Clinical Rheumatology 2010 5:5, 581-591
- [Background] Pincus T, Swearingen CJ, Bergman M, Yazici Y. RAPID3 (Routine Assessment of Patient Index Data 3), a rheumatoid arthritis index without formal joint counts for routine care: proposed severity categories compared to disease activity score and clinical disease activity index categories. J Rheumatol. 2008 Nov;35(11):2136-47. doi: 10.3899/jrheum.080182. Epub 2008 Sep 15. PMID 18793006